CLINICAL TRIAL: NCT04100707
Title: Efficacy of Genicular Nerve Radiofrequency in Patients With Knee Pain After Total Knee Replacement
Brief Title: Efficacy of Genicular Nerve Radiofrequency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Alp ALPTEKIN, University of Health Sciences, Diskapi Yildirim Beyazit Training and Research Hospital, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: diskapi01
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Chronic Pain
Keywords: Genicular nerve; Knee pain; Ultrasound
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operated (Experimental): Genicular block will aply to the patients with knee pain who was operated before
  Interventions: Procedure: Genicular block was applied
- Nonoperated (Sham Comparator): Genicular block will aply to the patients with knee pain who wasn't operated before
  Interventions: Procedure: Genicular block was applied

INTERVENTIONS:
Procedure: Genicular block was applied — This procedure is performed with ultrasound and / or fluoroscopy, sterile staining and covering of painful knee to the middle of thigh and leg, localization of superomedial, superolateral, inferomedial genicular nerves are tested and then conventional radiofrequency is applied to all 3 nerve regions

SUMMARY:
In patients with knee pain, local anesthetics and radiofrequency applications to superolateral, superomedial and inferomedial genicular nerves that innervate the knee joint are also preferred methods besides analgesic and physical therapy. When necessary, total knee replacement is the preferred method for primary knee arthrosis.

However, continuing knee pain is reported in approximately 20% of patients after total knee replacement. In similar cases; In the painful knees, the blockages of the genicular nerves are successfully applied.

In this study; the efficacy of imaging-guided radiofrequency application will be investigated in patients presenting with knee pain after total knee replacement.

DETAILED DESCRIPTION:
Although simple analgesic and physical therapy methods are applied, some patients suffer from pain. Genicular nerve blocks and radiofrequency methods are performed usually for this reason. This procedure is performed with ultrasound and / or fluoroscopy, sterile staining and covering of painful knee to the middle of thigh and leg, localization of superomedial, superolateral, inferomedial genicular nerves are tested and then conventional radiofrequency is applied to all 3 nerve regions.Fifty patients who had total knee prosthesis for gonarthrosis in the Orthopedics and Traumatology Clinic at least 3 months postoperatively had knee pain (infection, mechanical causes and radicular pain) were included in the study.The VAS and WOMAC values recorded at the time of application and the VAS and WOMAC values recorded at the 1st week, 1st month and 3rd month after the procedure will be used to evaluate the effectiveness of the method.

ELIGIBILITY:
Inclusion Criteria:

* knee pain

Exclusion Criteria:

* with communication problems (VAS and WOMAC scores could not be evaluated)
* infectious-mechanical pain-related conditions,
* with radicular pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-20 (Estimated); Primary Completion 2019-10-04 (Estimated); Study Completion 2019-11-04 (Estimated)

PRIMARY OUTCOMES:
Post intervention analgesic effect | at first 3 months
  Post intervention analgesic effects of genicular block on patients will be recorded. Postoperative pain, digital evaluation scale (Visual analogue scale -VAS; 0= absence of pain, 100= unbearable pain) of all patients will be performed and recorded.

SECONDARY OUTCOMES:
Ultrasound versus fluoroscopy | at first 3 months
  Western Ontario and Mc Masters Osteoarthritis index (VOMAC) will be used to evaluate functional status on the efficacy of Ultrasound and fluoroscopy use.VOMAC is a disease-specific score in which pain, stiffness and physical functions are evaluated. It consists of 24 questions, 5 of which are pain, 2 are stiffness and 17 are evaluating physical function. It has both total score and subgroups can be evaluated separately. Maximum scores were 20 for pain subgroup, 8 for stiffness and 68 for physical function. High scores indicate that the patient has poor values in that group.

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Teaching and Research Hospital, Ankara, Turkey (Türkiye)